CLINICAL TRIAL: NCT02513446
Title: Effect of Multiple Doses of Itraconazole on the Pharmacokinetics of a Single Oral Dose of BI 1026706 in Healthy Male Subjects (an Open-label, Randomised, Two-period, Two-sequence Crossover Study)
Brief Title: Effect of Multiple Doses of Itraconazole on the Pharmacokinetics of a Single Oral Dose of BI 1026706 in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1320.20; 2015-002140-14 (EudraCT Number: EudraCT)
Record Dates: First submitted 2015-07-30; First posted 2015-07-31 (Estimated); Results first posted 2019-03-29 (Actual); Last update posted 2019-03-29 (Actual); Status verified 2018-12

CONDITIONS: Healthy
MeSH Terms: interventions — Itraconazole

ARMS (2):
- BI 1026706 (Experimental): Single dose
  Interventions: Drug: BI 1026706
- BI 1026706 + Itraconazole (Experimental): 7 days of itraconazole treatment combined with a single dose of 1026706 on day 4
  Interventions: Drug: BI 1026706; Drug: Itraconazole

INTERVENTIONS:
Drug: BI 1026706 — Single dose of BI 1026706 on Day 1
Drug: Itraconazole — 7 days of itraconazole treatment combined with a single dose of BI 1026706 on the fourth day
  Arms: BI 1026706 + Itraconazole

SUMMARY:
The primary objective of this trial is to investigate the effect of multiple doses of itraconazole on the pharmacokinetics of BI 1026706 given as single dose. The assessment of safety and tolerability of BI 1026706 is an additional objective of this trial. Furthermore, the pharmacokinetics of the metabolite BI 1072668 will be explored.

ELIGIBILITY:
Inclusion criteria:

* Healthy male subjects according to the investigators assessment, based on a complete medical history including a physical examination, vital signs (BP, PR), 12-lead ECG, and clinical laboratory tests
* Age of 18 to 55 years (incl.)
* BMI of 18.5 to 29.9 kg/m2 (incl.)
* Signed and dated written informed consent prior to admission to the study in accordance with GCP and local legislation

Exclusion criteria:

* Any finding in the medical examination (including BP, PR or ECG) is deviating from normal and judged as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 50 to 90 bpm
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease judged as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy and simple hernia repair)
* Diseases of the central nervous system (such as epilepsy), other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Chronic or relevant acute infections
* History of relevant allergy or hypersensitivity (including allergy to the trial medication or its excipients)
* Intake of drugs with a long half-life (more than 24 h) within 30 days or less than 10 half-lives of the respective drug prior to administration of trial medication
* Within 10 days prior to administration of trial medication, use of drugs that might reasonably influence the results of the trial or that might prolong the QT/QTc interval
* Participation in another trial where an investigational drug has been administered within 60 days prior to planned administration of trial medication
* Smoker (more than 10 cigarettes or 3 cigars or 3 pipes per day)
* Inability to refrain from smoking during in-house confinement at trial site
* Alcohol abuse (consumption of more than 30 g per day)
* Drug abuse or positive drug screening
* Blood donation of more than 100 mL within 30 days prior to administration of trial medication or intended donation during the trial
* Intention to perform excessive physical activities within one week prior to administration of trial medication or during the trial
* Inability to comply with dietary regimen of trial site
* A marked baseline prolongation of QT/QTc interval (such as QTc intervals that are repeatedly greater than 450 ms) or any other relevant ECG finding at screening
* A history of additional risk factors for Torsades de Pointes (such as heart failure, hypokalaemia, or family history of Long QT Syndrome)
* Subject is assessed as unsuitable for inclusion by the investigator, for instance, because the subject is considered not able to understand and comply with study requirements, or because he has a condition that would not allow safe participation in the study

In addition, the following trial-specific exclusion criteria apply:

* Liver enzyme (ALT, AST, GGT) values above upper limit of normal at the screening examination
* Galactose intolerance, lactase deficiency, or glucose/galactose malabsorption

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2015-09-29 (Actual); Primary Completion 2015-11-14 (Actual); Study Completion 2015-11-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1320.20.1 Boehringer Ingelheim Investigational Site, Biberach, Germany

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: An open-label, randomised, two-period, two-sequence crossover study with healthy male subjects
Groups:
- Sequence RT: Treatment R (BI 1026706 alone):
  Oral administration of a single dose of 25 mg BI 1026706 film-coated tablets was given on Day 1.
  Treatment T (itraconazole + BI 1026706):
  Itraconazole (200 mg) as capsules was given orally twice daily as a loading dose on Day -3 and once daily from Day -2 to Day 4 (7 days in total). A single dose of 25 mg BI 1026706 was given orally on the fourth day (Day 1) of the itraconazole treatment (1 h after the itraconazole administration on the respective day).
  The single dose administrations of BI 1026706 in treatments R and T were separated by a wash-out period of at least 10 days.
- Sequence TR: Treatment T (itraconazole + BI 1026706):
  Itraconazole (200 mg) as capsules was given orally twice daily as a loading dose on Day -3 and once daily from Day -2 to Day 4 (7 days in total). A single dose of 25 mg BI 1026706 was given orally on the fourth day (Day 1) of the itraconazole treatment (1 h after the itraconazole administration on the respective day).
  Treatment R (BI 1026706 alone):
  Oral administration of a single dose of 25 mg BI 1026706 film-coated tablets was given on Day 1.
  The single dose administrations of BI 1026706 in treatments T and R were separated by a wash-out period of at least 10 days.
Period: Period 1
Arm/Group | Sequence RT | Sequence TR
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0
Period: Washout Period of 10 Days
Arm/Group | Sequence RT | Sequence TR
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0
Period: Period 2
Arm/Group | Sequence RT | Sequence TR
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): The TS included all subjects of the randomised set (RS), who were documented to have taken at least 1 dose of trial medication. It was used to assess safety, demographics, and other baseline characteristics as well as concomitant diseases and medications.
  The RS contained all entered (i.e. randomised) subjects.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sequence RT | Sequence TR | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.9 (10.2) | 33.0 (8.1) | 35.4 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 8 | 8 | 16

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve of BI 1026706 From 0 to the Last Quantifiable Data Point (AUC0-tz)
Description: Area under the concentration-time curve of BI 1026706 in plasma over the time interval from 0 to the last quantifiable data point (AUC0-tz)
Time Frame: -3 hours (h) before drug administration and 0.25h, 0.5h, 0.75h, 1h, 1.5h, 2h, 3h, 4h, 6h, 8h, 10h, 12h, 24h, 34h, 47h, 71h and 95h after drug administration
Population: Pharmacokinetic set (PKS) included all treated subjects that provided at least 1 primary or secondary pharmacokinetic parameter that was not excluded due to a protocol violation relevant to the evaluation of pharmacokinetics or due to pharmacokinetic non-evaluability..
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Groups:
- Treatment R (BI 1026706 Alone): Oral administration of single dose of 25 mg BI 1026706 was given on Day 1.
- Treatment T (Itraconazole + BI 1026706): Itraconazole (200 mg) was given orally twice daily as a loading dose on Day -3 and once daily from Day -2 to Day 4 (7 days in total). A single dose of 25 mg BI 1026706 was given orally on the fourth day (Day 1) of the itraconazole treatment (1 h after the itraconazole administration on the respective day).
Arm/Group | Treatment R (BI 1026706 Alone) | Treatment T (Itraconazole + BI 1026706)
Number analyzed (Participants) | 16 | 15
nmol*h/L | 921 (47.8) | 1580 (55.9)
Statistical Analysis 1: Comparison: Treatment R (BI 1026706 Alone) vs Treatment T (Itraconazole + BI 1026706); Test type: Superiority or Other; ANOVA; Analysis of variance (ANOVA) on the logarithmic scale; Fixed effects: sequence, period and treatment; Random effects: subjects within sequences; Adjusted gMean T/R ratio = 176.1, 90% CI 2-sided [160.5 to 193.2] — Ratio of the treatment adjusted geometric means (gMean) of (T) versus (R)

2. Primary Outcome: Maximum Concentration of BI 1026706 (Cmax)
Description: Maximum measured concentration of BI 1026706 in plasma (Cmax)
Time Frame: 0.25h, 0.5h, 0.75h, 1h, 1.5h, 2h, 3h, 4h, 6h, 8h, 10h, 12h, 24h, 34h, 47h, 71h and 95h after drug administration
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | Treatment R (BI 1026706 Alone) | Treatment T (Itraconazole + BI 1026706)
Number analyzed (Participants) | 16 | 15
nmol/L | 206 (48.9) | 279 (62.2)
Statistical Analysis 1: Comparison: Treatment R (BI 1026706 Alone) vs Treatment T (Itraconazole + BI 1026706); Test type: Superiority or Other; ANOVA; [statistical method as in outcome 1, analysis 1]; Adjusted gMean T/R ratio = 136.5, 90% CI 2-sided [109.9 to 169.4] — Ratio of the treatment adjusted geometric means (gMean) of (T) versus (R)

3. Secondary Outcome: Area Under the Curve of BI 1026706 From 0 Extrapolated to Infinity (AUC0-inf)
Description: Area under the concentration-time curve of BI 1026706 in plasma over the time interval from 0 extrapolated to infinity (AUC0-inf)
Time Frame: as for outcome 1
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | Treatment R (BI 1026706 Alone) | Treatment T (Itraconazole + BI 1026706)
Number analyzed (Participants) | 16 | 15
nmol*h/L | 943 (46.9) | 1600 (54.6)
Statistical Analysis 1: Comparison: Treatment R (BI 1026706 Alone) vs Treatment T (Itraconazole + BI 1026706); Test type: Superiority or Other; ANOVA; [statistical method as in outcome 1, analysis 1]; Adjusted gMean T/R ratio = 174.8, 90% CI 2-sided [159.1 to 192.0] — Ratio of the treatment adjusted geometric means (gMean) of (T) versus (R)

ADVERSE EVENTS:
Time Frame: From first drug administration through the residual effect period (REP) until the individual subject's end-of-trial; Up to 14 days
Groups:
- Total: Total
Arm/Group | Treatment R (BI 1026706 Alone) | Treatment T (Itraconazole + BI 1026706) | Total
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 3/16 | 4/16 | 5/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment R (BI 1026706 Alone) (N=16) | Treatment T (Itraconazole + BI 1026706) (N=16) | Total (N=16)
Nasopharyngitis (Infections and infestations) | 1 | 1 | 2
Headache (Nervous system disorders) | 1 | 2 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No